CLINICAL TRIAL: NCT00668863
Title: A Phase II Study Of Sunitinib In Combination With Irinotecan, L-leucovorin, And 5-Fluorouracil In Patients With Unresectable Or Metastatic Colorectal Cancer
Brief Title: Study Of Sunitinib With FOLFIRI In Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: A6181151
Record Dates: First submitted 2008-04-25; First posted 2008-04-29 (Estimated); Results first posted 2011-10-07 (Estimated); Last update posted 2011-10-17 (Estimated); Status verified 2011-10

CONDITIONS: Unresectable or Metastatic Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Leucovorin; Fluorouracil; Sunitinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 1 (Experimental)
  Interventions: Drug: FOLFIRI (The combination regimen of Irinotecan, l-Leucovorin and 5-Fluorouracil); Drug: Sunitinib

INTERVENTIONS:
Drug: FOLFIRI (The combination regimen of Irinotecan, l-Leucovorin and 5-Fluorouracil) — FOLFIRI treatment with Sunitinib on Day, Irinotecan 180M/M IV , l-Leucovorin 200M/M, 5FU 400M/M bolus and 2400M/M in 46-hour continuous infusion on Day1 each 42 day cycle. Number of Cycles: until progression or unacceptable toxicity develops.
Drug: Sunitinib — 37.5mg daily P.O., 4 weeks On 2weeks Off each 42 day cycle. Number of cycles: until progression or unacceptable toxicity develops.
  Other Names: Sutent

SUMMARY:
To evaluate the efficacy, safety and pharmacokinetics of sunitinib plus FOLFIRI (irinotecan, 5-FU and l-leucovorin) in the first-line treatment of Japanese mCRC patients

ELIGIBILITY:
Inclusion Criteria:

* Patient with histologically- or cytologically-confirmed colorectal adenocarcinoma with unresectable or metastatic disease documented on diagnostic imaging studies.
* Patient must have at least one RECIST-defined measurable lesion that has not been treated with prior local therapy.

Exclusion Criteria:

* History of another primary malignancy within 3 years prior to study entry, with the exception of non-melanoma skin cancer and in situ carcinoma of the uterine cervix.
* Current, recent, or planned participation in an experimental treatment drug study other than this protocol.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2008-05; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (10):
- Japan (10):
  - Pfizer Investigational Site, Nagoya, Aichi-ken
  - Pfizer Investigational Site, Chiba, Chiba
  - Pfizer Investigational Site, Matsuyama, Ehime
  - Pfizer Investigational Site, Sapporo, Hokkaido
  - Pfizer Investigational Site, Minoh/Osaka, Japan
  - Pfizer Investigational Site, Kochi, Kochi
  - Pfizer Investigational Site, Saku, Nagano
  - Pfizer Investigational Site, Osakasayama-shi, Osaka
  - Pfizer Investigational Site, Takatsuki, Osaka
  - Pfizer Investigational Site, Shimotsuke-shi, Tochigi

REFERENCES:
- [Derived] Tsuji Y, Satoh T, Tsuji A, Muro K, Yoshida M, Nishina T, Nagase M, Komatsu Y, Kato T, Miyata Y, Mizutani N, Hashigaki S, Lechuga MJ, Denda T. First-line sunitinib plus FOLFIRI in Japanese patients with unresectable/metastatic colorectal cancer: a phase II study. Cancer Sci. 2012 Aug;103(8):1502-7. doi: 10.1111/j.1349-7006.2012.02320.x. Epub 2012 Jun 14. PMID 22537162
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6181151&StudyName=Study%20Of%20Sunitinib%20With%20FOLFIRI%20In%20Colorectal%20Cancer

RESULTS

PARTICIPANT FLOW:
Groups:
- Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI: Sunitinib was orally administered at 37.5 mg once daily for 4 consecutive weeks followed by a 2-week rest period to comprise a complete cycle of 6 weeks (Schedule 4/2). Sunitinib was given in combination with FOLFIRI, which was administered in the standard fashion every 2 weeks: Irinotecan (180 mg/m^2) and l-leucovorin (200 mg/m^2) was infused intravenously on Day 1, immediately followed by 5 FU bolus (400 mg/m^2) and 46-hour (2400 mg/m^2) infusion. FOLFIRI was given on Days 1, 15, and 29 in each 6-week cycle of sunitinib administration.
Period: Overall Study
Arm/Group | Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI
Started | 71
Completed | 0
Not Completed | 71
Not completed — Objective Progression or Relapse | 42
Not completed — Adverse Event | 13
Not completed — Study Terminated by Sponsor | 8
Not completed — Global Deterioration of Health Status | 4
Not completed — Withdrawal by Subject | 1
Not completed — Surgery | 1
Not completed — Subject's work scheduling problem | 1
Not completed — Physician Decision | 1

BASELINE CHARACTERISTICS:
Arm/Group | Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI
Number analyzed (Participants) | 71
Age, Customized [Number; unit: participants]
  <=44 years | 6
  45 to 64 years | 44
  >=65 years | 21
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 29
  Male | 42

OUTCOME MEASURES:

1. Primary Outcome: Progression-Free Survival (PFS)
Description: PFS is defined as the time from the date of enrollment to the date of the first documentation of objective tumor progression or death due to any cause, whichever occurs first.
  PFS data was censored on the day following the date of the last tumor assessment documenting absence of progressive disease for patients who 1) were given anti-tumor treatment other than the study treatment prior to observing objective tumor progression; 2) were removed from the study prior to documentation of objective tumor progression; and 3) were ongoing at the time of the analysis.
Time Frame: Up to 11 cycles (1 cycle = 6 weeks)
Population: Full Analysis Set was defined as all enrolled subjects who met the following criteria :1) Those who were diagnosed as having adenocarcinoma of the colon or rectum with documented locally advanced or metastatic disease and 2) those who received at least one dose of the study medication.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI
Number analyzed (Participants) | 71
weeks | 28.9 [20.3 to 40.0]

2. Secondary Outcome: Overall Survival (OS)
Description: OS is defined as the time from the date of enrollment to the date of death due to any cause. OS data was censored on the day following the date of the last contact at which the patient is known to be alive.
Time Frame: Up to 11 cycles (1 cycle = 6 weeks)
Population: Median OS was not calculable due to the large number of censored events (63 out of 71 were censored).
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI
Number analyzed (Participants) | 0

3. Secondary Outcome: Percentage of Participants Who Presented Objective Response: Objective Response Rate (ORR)
Description: ORR is defined as the percentage of participants with best overall response of either a confirmed complete (CR) or partial response (PR) relative to the number of participants in FAS. Based on the response evaluation criteria in solid tumors (RECIST), CR is defined as the disappearance of all target lesions and PR is defined as a greater than or equal to 30% decrease in the sum of the longest dimensions of the target lesion.
Time Frame: Up to 11 cycles (1 cycle = 6 weeks)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: percentage of participants
Arm/Group | Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI
Number analyzed (Participants) | 71
percentage of participants | 36.6 [25.5 to 48.9]

4. Secondary Outcome: Duration of Response (DR)
Description: DR is defined as the time from the first objective documentation of complete or partial response that is subsequently confirmed to the first documentation of disease progression or to death due to any cause, whichever occurs first. The definition of censorship is the same as PFS.
Time Frame: Up to 11 cycles (1 cycle = 6 weeks)
Population: Analysis set was consisted of participants with a confirmed objective tumor response (CR or PR) among Full Analysis Set.
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI
Number analyzed (Participants) | 26
weeks | 28.3 [25.1 to 44.3]

5. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) and Predose Concentration (Ctrough) of Sunitinib.
Description: Plasma concentrations were assessed at predose, 2, 4, 6, 8, and 24 hours postdose and Cmax and Ctrough of sunitinib, its metabolite SU012662, and the total (sunitinib + SU0122662) were determined.
Time Frame: Cycle 1 Day 15
Population: Analysis set was consisted of participants who provided an evaluable sample. Planned number of participants for pharmacokinetic analysis was 6.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI
Number analyzed (Participants) | 3
ng/mL
  Sunitinib Cmax | 54.3 (6.54)
  Sunitinib Ctrough | 41.8 (16.4)
  SU012662 Cmax | 15.8 (3.96)
  SU012662 Ctrough | 11.3 (1.41)
  Total (sunitinib + SU0122662) Cmax | 70.0 (4.67)
  Total (sunitinib + SU0122662) Ctrough | 53.1 (15.4)

6. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Sunitinib
Time Frame: Cycle 1 Day 15
Population: as for outcome 5
Measure: Mean (Full Range); unit: hours
Arm/Group | Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI
Number analyzed (Participants) | 3
hours
  Sunitinib Tmax | 6 [0 to 8]
  SU012662 Tmax | 4 [4 to 8]
  Total (sunitinib + SU0122662) Tmax | 6 [4 to 8]

7. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 to 24 Hours Postdose (AUC 0-24) of Sunitinib
Description: AUC 0-24 was determined using the Linear/Log trapezoidal method.
Time Frame: Cycle 1 Day 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI
Number analyzed (Participants) | 3
ng.h/mL
  Sunitinib AUC 0-24 | 1161 (200)
  SU012662 AUC 0-24 | 346 (108)
  Total (sunitinib + SU0122662) AUC 0-24 | 1507 (114)

8. Secondary Outcome: Apparent Oral Clearance (CL/F) of Sunitinib
Description: Clearance of a drug is a measure of the rate at which a drug is metabolized or eliminated by normal biological processes. Clearance obtained after oral dose (apparent oral clearance) is influenced by the fraction of the dose absorbed. Clearance was estimated from population pharmacokinetic (PK) modeling. Drug clearance is a quantitative measure of the rate at which a drug substance is removed from the blood.
Time Frame: Cycle 1 Day 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI
Number analyzed (Participants) | 3
L/hour | 32.9 (6.25)

9. Secondary Outcome: Maximum Observed Plasma Concentration (Cmax) of Irinotecan
Description: Plasma samples were assessed at prior to initiation of irinotecan (and l-leucovorin) infusion, 1, 2 (predose for 5-FU bolus), 4, 8, and 24 hours after initiation of irinotecan infusion, and Cmax of irinotecan and its metabolite SN-38 were determined.
Time Frame: Cycle 1 Day 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI
Number analyzed (Participants) | 3
ng/mL
  Irinotecan Cmax | 1963 (492)
  SN-38 Cmax | 25.1 (7.29)

10. Secondary Outcome: Time to Reach Maximum Plasma Concentration (Tmax) of Irinotecan
Time Frame: Cycle 1 Day 15
Population: as for outcome 5
Measure: Mean (Full Range); unit: hours
Arm/Group | Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI
Number analyzed (Participants) | 3
hours
  Irinotecan tmax | 2 [1 to 2]
  SN-38 tmax | 4 [2 to 4]

11. Secondary Outcome: Area Under the Plasma Concentration Versus Time Curve From Time 0 to the Time of the Last Measurable Concentration (AUC Last) and Area Under the Plasma Concentration Versus Time Curve From Time 0 to Infinity (AUC ∞) of Irinotecan
Description: AUC last of irinotecan and its metabolite SN-38 were calculated using the Linear/Log trapezoidal method.
  AUC∞ of irinotecan was calculated using following equation; AUC last+(C*t/kel), where Ct* is the estimated concentration at the time of the last quantifiable concentration, kel is terminal phase rate constant that is estimated as the absolute value of the slope of a linear regression during the terminal phase of the natural-logarithm (ln) transformed concentration-time profile.
Time Frame: Cycle 1 Day 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng.h/mL
Arm/Group | Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI
Number analyzed (Participants) | 3
ng.h/mL
  Irinotecan AUC last | 13100 (1323)
  Irinotecan AUC ∞ | 13800 (1400)
  SN-38 AUC last | 274 (117)

12. Secondary Outcome: Terminal Phase Elimination Half-life (t1/2) of Irinotecan
Description: Terminal phase half-life of irinotecan was calculated as ln 2/ kel.
Time Frame: Cycle 1 Day 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI
Number analyzed (Participants) | 3
hours | 5.36 (0.221)

13. Secondary Outcome: Clearance of Irinotecan
Description: CL is calculated as dose divided by AUC 0-∞
Time Frame: Cycle 1 Day 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L/hour
Arm/Group | Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI
Number analyzed (Participants) | 3
L/hour | 23.0 (1.53)

14. Secondary Outcome: Volume of Distribution at Steady State (Vss) of Irinotecan
Description: Vss was calculated using following equation: CL x mean residence time (MRT), where MRT = the area under the first moment curve from zero time to infinity (AUMC 0-∞)/AUC 0-∞- (infusion time/2), AUMC 0-∞ = the area under the first moment curve from zero time to time t (AUMC t)+ ((t x Ct*)/ kel) + (Ct* / kel^2), AUMC t is calculated using the linear trapezoidal method.
Time Frame: Cycle 1 Day 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: L
Arm/Group | Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI
Number analyzed (Participants) | 3
L | 160 (16.8)

15. Secondary Outcome: Plasma Concentration at Steady State (Css) of 5-FU
Description: Concentration at 22 hour post start of 5-FU infusion were to be used as Css if 5-FU concentrations suggested steady state at 22 hours time point.
Time Frame: Cycle 1 Day 15
Population: as for outcome 5
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI
Number analyzed (Participants) | 3
ng/mL | 650 (70.5)

16. Secondary Outcome: Number of Participants With Adverse Events (AEs), Serious Adverse Events (SAEs), and Grade 3 or Higher Adverse Events According to Common Terminology Criteria (CTCAE).
Description: Any untoward medical occurrence in a patient who received study drug was considered an adverse event (AE), without regard to possibility of causal relationship. Treatment-emergent adverse events (TEAE): those which occurred or worsened after baseline. An adverse event resulting in any of the following outcomes, or deemed to be significant for any other reason, was considered to be a serious adverse event (SAE): death; initial or prolonged inpatient hospitalization; a life-threatening experience (immediate risk of dying); persistent or significant disability/incapacity; congenital anomaly.
Time Frame: Up to 11 cycles (1 cycle = 6 weeks)
Population: Safety analysis set was defined as the same population as the Full Analysis Set.
Measure: Number; unit: Participants
Arm/Group | Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI
Number analyzed (Participants) | 71
Participants
  Treatment emergent adverse events | 71
  Serious adverse events | 32
  CTCAE grade 3 or 4 adverse events | 70
  CTCAE grade 5 adverse events | 1

ADVERSE EVENTS:
Time Frame: Up to 11 cycles (1 cycle = 6 weeks)
Description: The same event may appear as both an AE and a SAE. However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Arm/Group | Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI
Serious Adverse Events (participants affected / at risk) | 32/71
Other Adverse Events (participants affected / at risk) | 71/71
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI (N=71)
Febrile neutropenia (Blood and lymphatic system disorders) | 6
Leukopenia (Blood and lymphatic system disorders) | 2
Lymphadenitis (Blood and lymphatic system disorders) | 1
Neutropenia (Blood and lymphatic system disorders) | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 2
Myocardial infarction (Cardiac disorders) | 1
Diarrhoea (Gastrointestinal disorders) | 1
Gastric dilatation (Gastrointestinal disorders) | 1
Gastrointestinal perforation (Gastrointestinal disorders) | 1
Haemorrhoids (Gastrointestinal disorders) | 1
Ileus (Gastrointestinal disorders) | 1
Intestinal obstruction (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 4
Pneumatosis intestinalis (Gastrointestinal disorders) | 1
Vomiting (Gastrointestinal disorders) | 5
Fatigue (General disorders) | 2
Pyrexia (General disorders) | 1
Abdominal abscess (Infections and infestations) | 1
Infection (Infections and infestations) | 1
Influenza (Infections and infestations) | 1
Localised infection (Infections and infestations) | 1
Pneumonia (Infections and infestations) | 1
Septic shock (Infections and infestations) | 1
Wound complication (Injury, poisoning and procedural complications) | 1
Wound dehiscence (Injury, poisoning and procedural complications) | 1
Neutrophil count decreased (Investigations) | 3
White blood cell count decreased (Investigations) | 1
Decreased appetite (Metabolism and nutrition disorders) | 6
Dehydration (Metabolism and nutrition disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Hydronephrosis (Renal and urinary disorders) | 1
Hypertension (Vascular disorders) | 1
Thrombosis (Vascular disorders) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Sunitinib 37.5 mg (Schedule 4/2) + FOLFIRI (N=71)
Anaemia (Blood and lymphatic system disorders) | 4
Febrile neutropenia (Blood and lymphatic system disorders) | 11
Leukopenia (Blood and lymphatic system disorders) | 4
Neutropenia (Blood and lymphatic system disorders) | 4
Thrombocytopenia (Blood and lymphatic system disorders) | 4
Hypothyroidism (Endocrine disorders) | 4
Eyelid oedema (Eye disorders) | 5
Abdominal distension (Gastrointestinal disorders) | 6
Abdominal pain (Gastrointestinal disorders) | 13
Abdominal pain upper (Gastrointestinal disorders) | 10
Cheilitis (Gastrointestinal disorders) | 8
Constipation (Gastrointestinal disorders) | 29
Diarrhoea (Gastrointestinal disorders) | 55
Dyspepsia (Gastrointestinal disorders) | 6
Gingivitis (Gastrointestinal disorders) | 13
Haemorrhoids (Gastrointestinal disorders) | 5
Nausea (Gastrointestinal disorders) | 54
Stomatitis (Gastrointestinal disorders) | 36
Vomiting (Gastrointestinal disorders) | 39
Face oedema (General disorders) | 8
Fatigue (General disorders) | 47
Malaise (General disorders) | 8
Mucosal inflammation (General disorders) | 9
Oedema (General disorders) | 6
Oedema peripheral (General disorders) | 6
Pyrexia (General disorders) | 27
Infection (Infections and infestations) | 5
Nasopharyngitis (Infections and infestations) | 12
Alanine aminotransferase increased (Investigations) | 18
Aspartate aminotransferase increased (Investigations) | 16
Blood albumin decreased (Investigations) | 22
Blood alkaline phosphatase increased (Investigations) | 13
Blood bilirubin increased (Investigations) | 7
Blood cholesterol increased (Investigations) | 5
Blood creatinine increased (Investigations) | 6
Blood glucose increased (Investigations) | 9
Blood lactate dehydrogenase increased (Investigations) | 5
Blood phosphorus decreased (Investigations) | 15
Blood potassium decreased (Investigations) | 5
Blood thyroid stimulating hormone increased (Investigations) | 4
Blood triglycerides increased (Investigations) | 4
C-reactive protein increased (Investigations) | 5
Gamma-glutamyltransferase increased (Investigations) | 11
Haemoglobin decreased (Investigations) | 28
Lymphocyte count decreased (Investigations) | 24
Neutrophil count decreased (Investigations) | 65
Platelet count decreased (Investigations) | 56
Protein total decreased (Investigations) | 6
Protein urine present (Investigations) | 7
Red blood cell count decreased (Investigations) | 4
Weight decreased (Investigations) | 7
White blood cell count decreased (Investigations) | 64
Decreased appetite (Metabolism and nutrition disorders) | 50
Dehydration (Metabolism and nutrition disorders) | 5
Diabetes mellitus (Metabolism and nutrition disorders) | 4
Back pain (Musculoskeletal and connective tissue disorders) | 11
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 5
Dizziness (Nervous system disorders) | 12
Dysgeusia (Nervous system disorders) | 35
Headache (Nervous system disorders) | 12
Neuropathy peripheral (Nervous system disorders) | 4
Insomnia (Psychiatric disorders) | 11
Proteinuria (Renal and urinary disorders) | 5
Cough (Respiratory, thoracic and mediastinal disorders) | 7
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 10
Hiccups (Respiratory, thoracic and mediastinal disorders) | 10
Alopecia (Skin and subcutaneous tissue disorders) | 44
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 33
Pruritus (Skin and subcutaneous tissue disorders) | 5
Rash (Skin and subcutaneous tissue disorders) | 12
Skin discolouration (Skin and subcutaneous tissue disorders) | 22
Flushing (Vascular disorders) | 4
Hypertension (Vascular disorders) | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.